CLINICAL TRIAL: NCT00236574
Title: A Randomized Double Blind Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Galantamine in Patients With Mild Cognitive Impairment (MCI) Clinically at Risk for Development of Clinically Probable Alzheimer's Disease.
Brief Title: A Study to Evaluate the Efficacy and Safety of Galantamine in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003145
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-11

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Dementia; Alzheimer disease; Mild cognitive impairment; Galantamine hydrobromide; Memory disorder
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction; Memory Disorders | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine hydrobromide

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of galantamine treatment in patients with mild cognitive impairment.

DETAILED DESCRIPTION:
This is an international, multicenter, double-blind, randomized, placebo-controlled trial. Following a 4 week screening period, patients with mild cognitive impairment (MCI), who are clinically at risk for development of Alzheimer's disease, will be randomized to treatment with either placebo or galantamine for 24 months with either placebo or a flexible dose of galantamine. Efficacy will be evaluated by measures of memory and cognition (Alzheimer's Disease Assessment Scale of cognition for MCI [ADAS-cog/MCI] and the Clinical Dementia Rating Sum of the Boxes [CDR-SB]), global severity of dementia (Clinical Dementia Rating [CDR]), functionality (Alzheimer's Disease Cooperative Study - Activities of Daily Living adapted to MCI [ADCS-ADL/MCI]), and changes on serial magnetic resonance imaging (MRI). Safety will be assessed using adverse event reports, vital signs, laboratory parameters, physical examination and electrocardiograms. The primary study hypothesis is that galantamine will improve memory deficits associated with mild cognitive impairment and therefore improve or stabilize the patient's cognitive abilities. A second study hypothesis is that treatment with galantamine slows or delays conversion of mild cognitive impairment to the dementia often associated with probable Alzheimer's disease in these patients. The third study hypothesis is that the treatment will be well tolerated by the patients. Galantamine hydrobromide immediate-release tablets (4, 8, and 12 milligrams (mg)) taken by mouth 2 times daily: 4 weeks at 8mg/day, 4 weeks at 16mg/day, increased to 24mg/day for the remainder of the 24-month trial. Dose may be reduced at investigator's discretion after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical decline of cognitive ability consistent with mild cognitive impairment
* Delayed recall score less than or equal to 10 on New York University paragraph recall test
* Sufficient visual, hearing and communication capabilities and willingness to complete serial standard tests of cognitive function
* Have a consistent informant to accompany them on scheduled visits
* Be able to read, write and fully understand the language of the cognitive scales used in the study

Exclusion Criteria:

* Contraindications for magnetic resonance imaging, for example, presence of pacemaker or presence of metal in high risk areas
* Neurodegenerative disorders such as Parkinson's disease
* Cognitive impairment resulting from acute cerebral trauma, hypoxic cerebral damage, vitamin deficiency states, infections such as meningitis or AIDS, or primary of metastatic cerebral neoplasia
* Significant endocrine or metabolic disease
* Mental retardation
* Women who are pregnant, nursing, or lacking adequate contraception

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2001-05; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Memory and cognition (ADAS-cog/MCI and CDR-SB scores) at 12 months and Global functional skills and the overall severity of dementia (the CDR-SB and the overall CDR) at 24 months.

SECONDARY OUTCOMES:
Brain atrophy assessed by MRI, Digit Symbol Coding, Alzheimer's Disease Cooperative Study-ADL scale(MCI version) at 24 months. Safety evaluations (adverse event reports, vital signs, laboratory tests, physical examination, electrocardiograms) throughout.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- [Derived] van de Pol LA, Korf ES, van der Flier WM, Brashear HR, Fox NC, Barkhof F, Scheltens P. Magnetic resonance imaging predictors of cognition in mild cognitive impairment. Arch Neurol. 2007 Jul;64(7):1023-8. doi: 10.1001/archneur.64.7.1023. PMID 17620494
- See also: A study to evaluate the efficacy and safety of galantamine in patients with mild cognitive impairment. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=504&filename=CR003145_CSR.pdf